CLINICAL TRIAL: NCT02000752
Title: Influence of Acupuncture in the Placental Expulsion Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI 36/2010
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-09

CONDITIONS: Placental Expulsion Time
Keywords: Labor; Acupuncture; Placental expulsion time; Postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): In the intervention group with real acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the point Ren Mai 6. This point is located on the anterior midline, between the umbilicus and the upper part of the pubic symphysis, at a distance of 0.3d from the umbilicus, being d the distance from the umbilicus to the upper part of the pubic symphysis. A sterilized steel needle of 0.25x40 mm is inserted in this point at 15-30 mm, depending on the adipose tissue of the woman.
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): Regarding to the control group with sham acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the placebo point with a sterilized 0.25x40 mm steel needle. The control point is located at the same horizontal level than the Ren Mai 6 point, but at 0.6d to the left of the anterior midline of the mother. In this case, the sterilized steel needle of 0.25x25 mm is inserted 15 mm into the tissue.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture
  Other Names: acupuncture needles
  Arms: Acupuncture
Device: Sham acupuncture — Sham point acupuncture
  Other Names: acupuncture needles
  Arms: Sham acupuncture

SUMMARY:
In this study, a single blind randomized trial is carried out in order to compare placental detachment times when Ren Mai 6 is stimulated and when a different placebo point is used. So, a lower detachment time is assumed to be related to a higher uterine contraction, and, therefore, a decrease in the hemorrhage postpartum. We focus on measuring the time it takes to placental delivery due to the fact that, if this point promotes the uterine contraction, then the placental delivery will be produced in a short time. Thus, this technique could decrease the hemorrhage postpartum.

The principal outcome of the study is the placental expulsion time. This time is measured by the midwife who is responsible of the birth, and it considers the time passed between the delivery of the newborn and the complete expulsion of the placenta.

Concerning the secondary outcomes, the application of real acupuncture in Ren Mai 6 point, and sham acupuncture in the placebo point are considered. Their study is derived from the statistical analysis of the results of the principal outcome. The existence of pain related to the treatment and the degree of satisfaction of the mother is also a secondary outcome, analyzed by the survey that the midwife carries out no more than 2 hours after the labor. At last, it is important to highlight that the degree of satisfaction of the midwife is also considered as a secondary outcome, since it is registered in the same survey.

DETAILED DESCRIPTION:
This study is designed as a single-blind randomized clinical trial with parallel design, and third party evaluation at the Hospital Universitario Príncipe de Asturias in Alcalá de Henares (Madrid, Spain). The study will be carry out with primiparous women who were in labour at this hospital. Information sheets about the study will be distributed by the different health care centers coordinated by the hospital. The midwives will give the information sheets to pregnant women during the pregnancy's attendances. The aim is to let pregnant women know about the study before their labour date in order to encourage them to participate in it.

Pregnant women fulfilling all the inclusion criteria and none of the exclusion criteria will be invited to participate in the experiment. These requirements includes primiparous women from 20 to 35 years old, with 37 to 42 weeks of gestation, and with a low obstetric risk labor with epidural analgesia. It is important to highlight that the midwife responsible for the labor is different from the acupuncturist responsible for the treatment.

An envelope with 120 leaflets will be enabled, 60 with control group name and 60 with intervention group name. After the approval of the pregnant woman, the acupuncturist will ask a partner midwife, a doctor or a nursing assistant to randomly pick up one of the leaflets from the aforementioned envelope, so pregnant woman will be assigned to a group. It is important to highlight that both the midwife and the pregnant woman must not know about the assigned group.

In the labor ward, after the childbirth, the baby is placed on the abdomen of the puerperal mother to facilitate maternal link. Then, the umbilical cord is clamped by the midwife. After all this process, that takes around a minute, the needle will be placed by the acupuncturist in the position corresponding to the randomly assigned group.

In the intervention group with real acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the point Ren Mai 6. This point is located on the anterior midline, between the umbilicus and the upper part of the pubic symphysis, at a distance of 0.3d from the umbilicus, being d the distance from the umbilicus to the upper part of the pubic symphysis. A sterilized steel needle of 0.25x40 mm will be inserted in this point at 15-30 mm, depending on the adipose tissue of the woman.

Regarding to the control group with sham acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the placebo point with a sterilized 0.25x40 mm steel needle. The control point is located at the same horizontal level than the Ren Mai 6 point, but at 0.6d to the left of the anterior midline of the mother. In this case, the sterilized steel needle of 0.25x25 mm will be inserted 15 mm into the tissue.

After the needle is punctured by the acupuncturist, the midwife waits for the placental expulsion, and pays attention on the time passed from the childbirth to the placental expulsion. After that, the time is registered into the partogram by the midwife. The needle will be then removed and the abdominal area completely sterilized by the acupuncturist.

A survey will be fulfilled by the midwife no more than 2 hours after the intervention. In this survey, the midwife takes notes on the comfort with which the technique was performed with four possible answers (high, moderate, medium and low comfort level). Furthermore, the acupuncturist will ask to the puerperal woman about the pain felt with the technique with four possible answers (painless, mild pain, moderate pain and high pain). The acupuncturist will also ask to the puerperal woman if she would recommend this technique to any of her friends with two possibles answers (yes or not).

Participants will be followed-up during the hospital stay, an expected average of 3 days. The expulsion placental time will be measured in the first thirty minutes after the childbirth is occurred. The satisfaction of professionals and participants, and the existence of pain during the technique will be registered into the 2 hours after the childbirth and before the puerperal woman is moved to the obstetrics plant which is out of the labor room. At last, the physician will annotate the existence of puerperal complications during the hospital stay in a specific sheet attached in the medical record of the woman. It will be done just before the woman discharges from the hospital, approximately three days after the labor.

In the medical record, an incidence form will be attached to be fulfilled in case of adverse events. So, the physician in charge of evaluating the welfare of the puerperal woman will register any kind of complication if it would have appeared. In other case, the physician will note the lack of complications.

Concerning the procedure and data collection, the acupuncturist will request permission to midwife responsible of the mother for their collaboration in the study in the pre-labor room. The acupuncturist will explain the study to the mother and her partner and will apply for her voluntary participation being the informed consent offered then. All information will be given when the pregnant woman is without pain of labor, preferably when the woman is under the epidural analgesia effects.

All the study will be performed in conditions of respect for individual rights and ethical principles affecting biomedical research involving human. Written informed consent will be fulfilled by all participants.

In particular, the physical and mental integrity of women will be safeguarded, as well as privacy and data protection in accordance to the spanish Organic Law 15/1999, of December 13, Protection of Personal Data. All the participants will give their informed consent in accordance with the Declaration of Helsinki (25) assuring confidentiality and freedom to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women between 20 and 35 years old
* Within 37 and 42 weeks of gestation
* Low obstetric risk labor
* With epidural analgesia

Exclusion Criteria:

* Myomatosis
* Coagulation disorders
* Placental alterations (placenta previa or placenta accreta)
* Uterine overdistension (multiple pregnancy, polyhydramnios or fetal macrosomia)
* Previous abortions and subject to curettage evacuator.
* Previous uterine surgeries
* Prolonged labor (more than 11 hours) or too fast labor (less than 2 hours)
* Use of uterine relaxants during childbirth (magnesium sulfate or halogenates anaesthetic drugs)
* People uncapable to give the informed consent

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Lopez Garrido, Midwife, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (1):
- Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three midwives responsible for conducting the study were trained in the acupuncture technique during a 3 hour seminar. None of the 3 acupuncture-trained midwives were responsible for the management of labor, birth, or the third stage of labor. The midwife responsible for the birth measured the duration of the third stage of labor in minutes.
Pre-assignment Details: Inclusion criteria included: primiparous, aged between 20 and 35 years, at 37 to 42 weeks gestation with a low risk labor, receiving epidural analgesia. All criteria were chosen to homogenize the sample and minimize the number of excluded women.
Groups:
- Acupuncture: In the intervention group with real acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the point Ren Mai 6. This point is located on the anterior midline, between the umbilicus and the upper part of the pubic symphysis, at a distance of 0.3d from the umbilicus, being d the distance from the umbilicus to the upper part of the pubic symphysis. A sterilized steel needle of 0.25x40 mm is inserted in this point at 15-30 mm, depending on the adipose tissue of the woman.
  Acupuncture
Period: Overall Study
Arm/Group | Sham Acupuncture | Acupuncture
Started | 60 | 60
Completed | 29 | 47
Not Completed | 31 | 13
Not completed — Dystocic delivery | 19 | 8
Not completed — Shift Changes | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 47 | 29 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.39 (4.95) | 29.38 (4.91) | 30.00 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 29 | 76
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 47 | 29 | 76

OUTCOME MEASURES:

1. Primary Outcome: The Principal Outcome of the Study is the Placental Expulsion Time.
Description: This time is measured by the midwife who is responsible of the birth, and it considers the time passed between the delivery of the newborn and the complete expulsion of the placenta.
Time Frame: Up to 30 minutes after the newborn delivery
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sham Acupuncture | Acupuncture
Number analyzed (Participants) | 29 | 47
minutes | 15.21 [12.70 to 17.71] | 5.23 [4.69 to 5.82]
Statistical Analysis 1: Comparison: Sham Acupuncture vs Acupuncture; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 9.98, 95% CI 1-sided [lower limit 7.59]

2. Secondary Outcome: Percentage of Participants Who Reported Experiencing Pain Related to Treatment
Description: The existence of pain related to the treatment is analyzed by the survey that the midwife carries out no more than 2 hours after the labor. A scale with 4 levels was used (no pain, mild pain, moderate pain, great pain).
Time Frame: Measured into the 2 hours after the childbirth but before puerperal woman is moved to the obstetrics plant out of the labor room
Measure: Number; unit: percentage
Arm/Group | Sham Acupuncture | Acupuncture
Number analyzed (Participants) | 29 | 47
percentage | 0 | 0
Statistical Analysis 1: Comparison: Sham Acupuncture vs Acupuncture; Test type: Superiority or Other; p = 1, t-test, 2 sided; difference in percentage = 0

3. Secondary Outcome: Percentage of Mothers That Would Recommend the Technique to Any of Her Friends
Description: The number of mothers that would recommend the technique to any of her friends is analyzed in the survey that the midwife carries out no more than 2 hours after the labor. The possible responses are "I would recommend it", or "I would not recommend it".
Time Frame: as for outcome 2
Measure: Number; unit: percentage
Arm/Group | Sham Acupuncture | Acupuncture
Number analyzed (Participants) | 29 | 47
percentage | 100 | 97.87
Statistical Analysis 1: Comparison: Sham Acupuncture vs Acupuncture; Test type: Superiority or Other; p = 0.16, t-test, 1 sided; difference in percentages = 2.13, 95% CI 1-sided [lower limit 1.01]

4. Secondary Outcome: Degree of Ease With Which the Acupuncturist Administered the Treatment
Description: The degree of ease with which the acupuncturist administered the treatment was measured in a survey that the midwife carries out no more than 2 hours after the labor. The value was recorded using a numerical scale ranging between 0-100, with 4 levels: "100 - high ease", "75 - moderate ease", "50 - medium ease" and "25 - low ease"
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Acupuncture | Acupuncture
Number analyzed (Participants) | 29 | 47
units on a scale | 93.97 (16.94) | 96.81 (8.34)
Statistical Analysis 1: Comparison: Sham Acupuncture vs Acupuncture; Test type: Superiority or Other; p = 0.2, t-test, 2 sided; Mean Difference (Final Values) = 2.84, 95% CI 1-sided [lower limit 0.84]

ADVERSE EVENTS:
Arm/Group | Sham Acupuncture | Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/47
Other Adverse Events (participants affected / at risk) | 0/29 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No